CLINICAL TRIAL: NCT06299969
Title: Feedback Intervention and Treatment Trial in Patients With Out-of-Hospital Cardiac Arrest (FITT-OHCA)
Brief Title: Feedback Intervention and Treatment Trial in Patients With Out-of-Hospital Cardiac Arrest
Acronym: FITT-OHCA
Status: Recruiting | Type: Observational
Sponsor: St.Bernward Hospital (Other)
Collaborators: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Karl Heinrich Scholz, Professor, St.Bernward Hospital
Other Study IDs: StBernwardH
Record Dates: First submitted 2023-12-29; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: OHCA; Out-of-hospital cardiac arrest; In-hospital cardiac arrest; Resuscitation; Cardiac arrest center; Feedback intervention; Acute care medicine
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The trial collects and analyzes data from Cardiac Arrest Centres in patients with out-of-hospital cardiac arrest (OHCA).

DETAILED DESCRIPTION:
With around 70,000 cases per year, out-of-hospital cardiac arrest (OHCA) is one of the most common causes of death in Germany. Only less than 10% of patients with an OHCA can currently be discharged with a satisfactory neurological outcome. The FITT-OHCA trial is a quality management project and collects data from Cardiac Arrest Centres on pre-hospital care and early post-resuscitation treatment in a standardized manner. The aim is to optimize the treatment process in patients following successful prehospital resuscitation through systematic data collection and feedback to the members of the rescue and treatment chain. The study includes cluster randomization of the participating hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients after cardiac arrest

Exclusion Criteria:

* refused register participation by patient or legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated after out-of-hospital cardiac arrest
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 3 weeks
  Death/Survival at discharge

SECONDARY OUTCOMES:
CPC score | 3 weeks
  Cerebral performance category
MRS | 3 weeks
  Modified ranking scale

CONTACTS AND LOCATIONS:
Locations (1):
- St Bernward Hospital, Hildesheim, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided